CLINICAL TRIAL: NCT02965222
Title: A Study Select Top-grade Embryo by Time-lapse Imaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WY710628
Record Dates: First submitted 2016-11-09; First posted 2016-11-16 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Top-grade Embryo
Keywords: blastocyst; pregnancy rate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention arm (Experimental): After injecting HCG 38- 40 hours , the patient's oocytes will be taken with ICSI , then placed in the Time-Lapse. The oocytes will be IVF after 4 hours and will be stripped surrounding cumulus cell ,then will be placed in the Time-Lapse.The third day the top-grade embryo will be selected by time-lapse imaging (TLI) . The cleavage pattern and time parameters for marker embryo development were recorded daily after insemination.
  Interventions: Device: the time-lapse videography
- Control arm (Experimental): The development of the embryos at time-lapse was recorded directly and was not disturbed by temperature changes.
  Interventions: Device: the time-lapse videography

INTERVENTIONS:
Device: the time-lapse videography — The all oocytes will be placed in the Time-Lapes .The third day the top-grade embryo will be selected by time-lapse imaging (TLI) .

SUMMARY:
To establish embryo time-difference kinetics scoring model for embryo selection before embryo transfer. It is especially suitable for selective single embryo transfer, advanced infertile women, and patients with repeated transplant failure. It can effectively improve clinical pregnancy rate, improve embryo implantation rate and Rate of return home. Reduce the risk of multiple pregnancies.

DETAILED DESCRIPTION:
1. BACKGROUND:

   At present, embryo selection in embryonic laboratories at various reproductive centers continues to follow conventional morphological assessments based on the time period provided by the 2016 Expert Consensus Guidelines for Laboratory Operations (revised from the Istanbul consensus) (discussion board), after insemination of the 1th-6th day (except the 4th day) to observe the specific time points of embryonic morphology, static observation, score, select the embryo. This method of observation of embryonic development is not comprehensive enough, and the lack of quantifiable recognized indicators .

   EmbryoScope Time-lapse culture system is the latest development of human assisted reproductive embryo from fertilization to blastocyst development. The time-lapse imaging system (TLI) is used to record the embryonic development process from fertilization to blastocyst formation. The timing of change plays a key role in the developmental potential of the embryo, such as the time of emergence and disappearance of pronucleus, the time of early cleavage, cleavage pattern and so on. At present, the latest 2016 Laboratory Operation Expert Consensus Guide (discussion board) provides a grading standard that does not objectively reflect specific information on morphological changes, such as cleavage patterns, the specific time of morphological changes, and so on for embryonic development and post- Determine the fate of embryos play a vital role. Due to the clinical diagnosis and treatment of the center of the standard, laboratory culture system, and the difference between the laboratory standard operation procedure,and embryonic development speed differences. Therefore, it is desirable to use the EmbryoScope Time-lapse culture system to find out the best timing of morphological changes of embryos in accordance with the laboratory culture system on the basis of the expert consensus time period. To establish an evaluation model of embryo morphology kinetics suitable for our laboratory. Embryology time-of-flight monitoring Morphological kinetics evaluation model is suitable for patients with in vitro fertilization/ intracytoplasmic sperm injection , especially for infertile women in assisted reproduction, women with repeated transplantation failure, women with fertility disorders requiring egg activation, Single embryo transfer of patients, effectively avoid multiple pregnancy, reduce the risk of multiple pregnancy. Selection of embryos with developmental potential for transplantation, improve embryo quality, improve the accuracy of embryo selection, contribute to successful pregnancy. But also can alleviate this part of the patient's mental stress, but also contribute to successful pregnancy. At the same time, for laboratory embryologists to provide more data reference, more human embryonic development information.

   At present, several large-scale centers are undergoing their own embryo laboratory kinetics of the scoring model. Shanshan Wang et al suggested that the cleavage pattern of embryos and time parameters combined to establish a new embryo screening model for single embryo transfer embryo, to obtain an ideal pregnancy outcome.

   EmbryoScope Time-lapse culture system and embryo selection, compared to the traditional culture system and the static morphology of the embryo selection, EmbryoScope Timelapse selection of transplanted embryos, the clinical pregnancy rate [3], EmbryoScope Time-lapse culture system, Significantly improved. The literature of N. Basile and P. Vime [4] suggests that blastocyst culture [10] plus the choice of embryo morphology kinetics may be the best treatment for improving clinical outcomes. Studies have been reported , time difference imaging system does not interfere with embryonic culture conditions in the case of interval 20 min, 5 min or 1 min to shoot images, and continued to the first 3 days or 5 days. In addition, the TLI image acquisition system can exclude some of the abnormal cleaved embryos that are considered to have "normal" developmental potential in static assessment. A number of studies have shown that the TLI culture system combined with the morphological scoring method to select the embryos obtained after transplantation compared with the purely morphological method of the choice of static embryos can be more satisfactory to patients with pregnancy outcomes .

   In this study, we compared the clinical outcomes of patients with two different culture routes, analyzed the advantages of TLI combined with morphological scoring methods, and established the model of embryonic time difference morphology kinetics in our laboratory. The aim of this study was to prospectively select embryos for selective single embryo transfer, advanced infertility women and patients with repeated graft failure to improve the clinical pregnancy rate and reduce the occurrence of multiple births.
2. Trial design:

   Samples were selected according to the inclusion criteria, and groups A and B were grouped according to the random number table, with 40-50 patients in each group. The random number table is attached. In order to avoid the withdrawal of patients or other reasons not suitable for inclusion in the trial, the researchers increased the sample size, the random number table increased to 150. A group of patients with oocytes injecting human chorionic gonadotrophin (HCG) 38-40 hours intracytoplasmic sperm injection (ICSI), and then into the ordinary three-gas incubator, conventional fertilization 4hours ,the demolition of eggs into the ordinary three-chamber, after insemination .The embryos were evaluated and selected by the current morphological scoring method. The oocytes of Group B were taken ICSI after infecting HCG 38-40 hours . And then be placed in the Time-Lapse. The ovaries were placed in the Time-Lapse after 4Hhours fertilization, and the embryos were evaluated by time-lapse imaging (TLI). The cleavage pattern and time parameters for marker embryo development were recorded daily after insemination. (1) The rate of high-quality embryos (cleavage and blastocyst stage), clinical pregnancy rate and embryo implantation rate in group A and group B; (2) The cleavage pattern and time parameters of embryo in group B were analyzed retrospectively, And the quality of blastocysts were analyzed. Logistic regression analysis was used to establish the criteria of embryo selection.

   (Age> 38 years), patients with recurrent graft failure (number of cycles ≥ 3), the development of embryos in this part of the patients were observed by TLI.Results: (1) Embryonic development , Select high-quality embryos for transplantation, observation of pregnancy outcome.
3. Statistical methods: The data were expressed as mean ± standard deviation (x ± s) or rate (%), and the data were analyzed by Statistical Package for the Social Sciences 23.0 software. The quartile method was used to classify the time parameters, and the advantage period of each parameter was calculated with the outcome of pregnancy and high quality blastocyst formation. Logistic regression analysis of clinical variables (cleavage patterns and time parameters) and the relationship between high-quality blastocysts, the rate of each group were compared using χ 2 test, P <0.05 for the difference was statistically significant.
4. Quality control and quality assurance Patients will managed by the listed investigators who have adequate experience in managing assisted reproduction treatments.A Trial steering committee will be formed which will oversee the conduct of the trial.
5. Data Handing and record keeping All data will be stored for three years. A desighnted research nurse will be responsible for data management including data coding,monitoring and verification.

ELIGIBILITY:
Inclusion Criteria:

1. women under 38 years of age
2. ≤2th cycle
3. transplantation cycle

Exclusion Criteria:

1. women with abnormal oocytes in the past(≥30%)
2. women with other systemic diseases
3. women with abnormal uterine cavity shown on hysterosalpingogram or saline infusion sonogram

Max Age: 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
live birth rate | 1 year
  numer of live birth per transfer cycle

SECONDARY OUTCOMES:
clinical pregnancy rate | 1year
implantation rate | 1year

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai first Maternity and Infant health hospital, Tong Ji University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Basile N, Vime P, Florensa M, Aparicio Ruiz B, Garcia Velasco JA, Remohi J, Meseguer M. The use of morphokinetics as a predictor of implantation: a multicentric study to define and validate an algorithm for embryo selection. Hum Reprod. 2015 Feb;30(2):276-83. doi: 10.1093/humrep/deu331. Epub 2014 Dec 19. PMID 25527613
- [Background] Rubio I, Galan A, Larreategui Z, Ayerdi F, Bellver J, Herrero J, Meseguer M. Clinical validation of embryo culture and selection by morphokinetic analysis: a randomized, controlled trial of the EmbryoScope. Fertil Steril. 2014 Nov;102(5):1287-1294.e5. doi: 10.1016/j.fertnstert.2014.07.738. Epub 2014 Sep 11. PMID 25217875
- [Background] Payne D, Flaherty SP, Barry MF, Matthews CD. Preliminary observations on polar body extrusion and pronuclear formation in human oocytes using time-lapse video cinematography. Hum Reprod. 1997 Mar;12(3):532-41. doi: 10.1093/humrep/12.3.532. PMID 9130755